CLINICAL TRIAL: NCT05646550
Title: Phase I Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of the Bispecific Antibody CC-1 in Men With Biochemical Recurrence of Prostate Cancer
Brief Title: Antibody CC-1 in Men With Biochemical Recurrence of Prostate Cancer
Acronym: ProSperACC-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ProSperA_CC-1; 2022-002420-13 (EudraCT Number); 2024-511430-12-00 (EU CTIS Number)
Record Dates: First submitted 2022-09-27; First posted 2022-12-12 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer Recurrent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Part (Experimental): In the dose escalation part, up to 7 dose cohorts will be included depending on occurrence of dose-limiting toxicity (DLT). Each dose cohort has a predefined day 3 dose level (DL): cohort 1, 78µg; cohort 2, 110µg; cohort 3, 150µg; cohort 4, 210µg; cohort 5, 300µg; cohort 6, 400µg; cohort 7, 600µg. Each dose cohort will consist of at least three patients evaluable for DLT. Maximum tolerated dose (MTD) is defined on at least six patients
  Interventions: Drug: CC-1 Infusion
- Dose Expansion Part (Experimental): CC-1 is administered as a 3-hour short-term intravenous infusion started at the MTD dose level identified in the dose escalation part of the study or based on the discretion of the sponsors delegate and DSMB recommendation supported by preliminary safety and efficacy data to constitute a modified MTD, e.g. to be one or more dose levels lower than the MTD determined. Patients can be treated simultaneously during the dose expansion phase. Patients must be hospitalized during step dosing, i.e. from day 1-4 (last dosing on day 3) of the first cycle. Thereafter inpatient treatment (overnight stay) depends on the discretion of the investigator, an outpatient treatment is preferred.
  Interventions: Drug: CC-1 Infusion

INTERVENTIONS:
Drug: CC-1 Infusion — Short term (3h) infusion of CC-1

SUMMARY:
This trial is a phase I open-label, single center study designed to evaluate the safety, tolerability and preliminary efficacy of the bispecific prostate specific membrane antigen (PSMA) and cluster of differentiation protein 3 (CD3) antibody CC-1 in men with biochemical recurrence (BCR) of prostate cancer (PC). The PSMA binder in CC-1 reacts with tumor cells and also binds to tumor vessels, thereby allowing for a dual mode of anti-cancer action. CC-1 was developed in a novel format, which not only prolongs serum half-life, but most importantly reduces off-target T-cell activation with accordingly reduced side effects. The study entails a part I (dose escalation part) to identify the maximally tolerated dose of CC-1, which then will be further evaluated in part II of the study (dose expansion part). After application of two low doses as safety steps in the first cycle, CC-1 will be applied twice weekly for three consecutive weeks within 4 week cycles as a short-term intravenous infusion (3 hours). The planned trial ultimately shall define the recommended phase II dose (RP2D) of CC-1 in the disease setting of BCR of PC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patient is able to understand and comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
* Men aged 18 and above
* Earlier histologic diagnosis of prostatic adenocarcinoma
* Low risk of rapid disease progression, defined as:

  - PSA-detection Time (DT) > 1 year AND pathological International Society of Urological Pathology (ISUP) grade < 4 for men with prior radical prostatectomy or Interval to biochemical recurrence > 18 months and biopsy ISUP grade < 4 for men with prior radiation therapy
* Biochemical recurrence (BCR) in compliance with the following 3 conditions:

  * after having finished last definitive treatment
  * PSA ≥0.2 ng/mL or PSA > nadir + 2 ng/mL (after definitive RT), with two increasing PSA values prior to study treatment
  * no distant metastasis upon PSMA- positron emission tomography (PET) imaging
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Male patients with partners of child-bearing potential, who are sexually active, must agree to the use of one highly effective form of contraception and one barrier method. This should be started from the signing of the informed consent and continue throughout period of taking study treatment and for 4 months after the last dose of study drug
* Adequate bone marrow, renal, and hepatic function defined by laboratory tests within 21 days prior to study treatment:

  * Hemoglobin ≥ 9 g/dl (Transfusion of packed red blood cells prior to enrolment allowed)
  * Neutrophil count ≥ 1,500/mm3
  * Platelet count ≥ 100,000/µl
  * Bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
  * gamma-glutamyl-transferase (γ-GT) ≤ 2.5 x ULN
  * prothrombin time (PT) - international normalised ratio (INR) / partial thromboplastin time (PTT) ≤ 1.5 x ULN
  * Creatine kinase ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 60 ml/min

Exclusion Criteria:

* PSA >5 ng/ml.
* For men with prior radical prostatectomy:

  * PSA-DT < 1 year or
  * pathological ISUP grade 4-5
* For men with prior radiation therapy:

  * Interval to biochemical recurrence < 18 months or
  * biopsy ISUP grade 4-5
* Other malignancy within the last 2 years except: adequately treated non-melanoma skin cancer and low-grade non-muscle invasive papillary bladder cancer.
* Concurrent or previous treatment within 30 days in another interventional clinical trial with an investigational anticancer therapy
* Patients who are receiving androgen-deprivation therapy.
* Patients who have received prior Androgen Deprivation Therapy (ADT) are not eligible with the exception of those that received ADT ≤ 36 months in duration and ≥9 months before enrolment and administered only in the neoadjuvant/adjuvant setting.
* Castrate level of serum testosterone <50 ng/dL at screening.
* History of HIV infection
* Viral active or chronic hepatitis (HBV or HCV)
* Ongoing autoimmune disease
* Current relevant central nervous system pathology (e.g. seizure, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder)
* Therapeutic anticoagulation
* Non-controlled hypertension, defined as mean blood pressure values in 24-hours blood pressure measurement of >130 mmHg or >90 mmHg for systolic or diastolic, respectively
* Heart failure defined as New York Heart Association (NYHA) III/IV
* Severe obstructive or restrictive ventilation disorder
* Known intolerance to CC-1 or other immunoglobulin drug products as well as hypersensitivity to any of the excipients present in CC-1

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose escalation part: To define the maximum tolerated dose (MTD) of CC-1 as 3 hours infusion | during the procedure
  Data Safety and Monitoring Board (DSMB) and Sponsor meeting about determination of the MTD for each cohort and the dose expansion phase
Dose expansion part: To define the recommended phase-II dose of CC-1 | up to 1 month after procedure
  Data Safety and Monitoring Board and Sponsor meeting about determination of the recommended phase II dose of CC-1 for potential phase II trials.

SECONDARY OUTCOMES:
To evaluate safety and tolerability of CC-1 | during the procedure
  Number of participants with Adverse Events (AEs) and with abnormal laboratory test results
To assess efficacy in terms of Prostata-Specific-Antigen (PSA) response and no PSA progression after CC-1 treatment | during the procedure and through study completion, an average of 6 months
  PSA response will be defined as ≥50% PSA decrease. In addition, "No PSA doubling", defined as PSA measured at visits C1-6, End Of Treatment (EOT), End Of Safety follow up (EOSf) and Follow-up (FU)1-5 divided by PSA measured at baseline, will be assessed as further efficacy endpoint. Furthermore, percentage of patients with no clinical relapse, no salvage and no subsequent antineoplastic therapy will be assessed
To assess clinical outcome in terms of progression-free survival, treatment-free survival, overall survival | through study completion, an average of 6 months
  Overall and progression free survival status as percentage of patients alive at EOSf and each follow-up assessment
To assess CC-1 serum concentrations | during the procedure prior to and after start of infusion on each treatment day in the first cycle (each cycle is 28 days).
  CC-1 serum concentrations assessed prior to and after start of infusion on each treatment day in the first cycle (each cycle is 28 days).
To assess quality of life | through study completion, an average of 1 year
  Quality of life is defined as overall quality of life scores European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ).

OTHER OUTCOMES:
To identify predictive biomarkers of response and resistance | during the procedure
  Samples for human anti-human antibody (HAHA) analysis
To evaluate pharmacokinetics and pharmacodynamics of CC-1 using Cytokine levels | baseline and immediately after procedure
  Cytokine levels in serum as assessed at baseline and after therapy using a commercially available, flow cytometry-based assay that allows parallel determination of different cytokines in one serum sample.

CONTACTS AND LOCATIONS:
Overall Officials: Walz, Prof. Dr., Principal Investigator — CCU Translational Immunology
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared with other researchers